CLINICAL TRIAL: NCT02471365
Title: NIEHS EPA Pilot Study of Exposure to Chemicals in Consumer Products
Brief Title: Study of Exposure to Chemicals in Consumer Products
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150134; 15-E-0134
Record Dates: First submitted 2015-06-12; First posted 2015-06-15 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-04-09

CONDITIONS: Product Use
Keywords: Exposure Assessment; Questionnaire; Product Use; Biomonitoring; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Non-pregnant and non-nursing females between 35 and 74 who usesa high number (e.g., 15 or more products a day) of consumer products.

SUMMARY:
Background:

- In a lifetime, a person may encounter tens of thousands of chemicals used as ingredients in the products they buy. It s not easy to measure them because the companies that sell the products don t have to tell the exact chemical ingredients. Researchers want to compare how existing methods (e.g., surveys and models) measure exposure to chemicals in personal care and household products.

Objective:

- To test and improve the ways that studies gather data about contact with chemicals found in consumer products.

Eligibility:

- Healthy women volunteers ages 35 74 who use at least 15 consumer products a day.

Design:

* Participants will be screened with medical history, pregnancy test, smoking test, and blood sample. They will answer questions about their homes and products they use.
* Participation will last about 30 hours over 12 days.
* Researchers will:
* Place air samplers inside and outside participants homes for 10 days. One sampler will need to be plugged into an electrical outlet. It will make a low, continuous sound while in operation.
* Collect house dust samples and record all consumer products in the house.
* Visit the house daily to collect samples.
* Participants will:
* Give a blood sample at a clinic twice.
* Collect all urine voids for 10 days. They will label it and put it in a special cooler.
* Wear 4 small devices that measure air pollution, chemicals, location, and activity.
* Record what they eat and what consumer products they use. They will write these in a diary and <TAB>photograph them on an iPhone provided to them.
* On day 2 of the study, they will collect a duplicate sample of what they eat.
* Take iPhone videos of their use of certain products.
* Answer questions about chemical ingredients in their personal care products.

DETAILED DESCRIPTION:
Research to advance the characterization of environmental and chemical exposures through improved exposure assessments, at both the individual and population levels, is a research priority identified in the Strategic Research Action Plan for the U.S. Environmental Protection Agency (EPA) s Chemical Safety for Sustainability (CSS) program (EPA 2012) and the National Institutes of Environmental Health Sciences (NIEHS) Strategic Plan for 2012-2017 (NIEHS 2012). Leading up to the Strategic Plan, specific research priorities related to exposure assessment were identified in the 2011 NIEHS workshop Advancing Research on Mixtures: New Perspectives and Approaches for Predicting Adverse Human Health Effects",

including the need to evaluate the utility of existing instruments that classify or quantify exposures, develop better tools to improve exposure assessment, and to better understand the nature of combined exposures (e.g., mixtures). This project will inform research priorities identified in the NIEHS strategic plan and several specific research needs discussed during the 2011 NIEHS workshop on mixtures, with a focus on assessing exposures from personal care and household products:

* Evaluate current exposure assessment technologies, including questionnaires
* Develop better models that link source with behavior to predict exposure
* Analyze combined exposures
* Evaluate usefulness of commercially available product use/marketing databases
* Evaluate prediction models
* Characterize behavior that impact exposures using new technologies (iPad/internet use)

Personal care products (PCPs) and other household/consumer products are of particular interest because of the efficiency of their delivery and widespread use. Exposure to chemicals in PCPs can result through either direct or indirect routes of contact depending on the use of the product (Dodson 2012; Koniecki et al. 2011; Rudel et al. 2003; Schettler 2006; Weschler and Nazaroff 2014). Health concerns exist about some chemicals found in PCPs and household setting. Over the course of a lifetime, the average consumer may encounter tens of thousands of chemicals used as ingredients in consumer products, many of which are proprietary; thus, getting a complete picture of the human exposome is challenging. Given the large number of co-occurring chemicals in these products, new strategies, tools, and

techniques need to be developed and evaluated for their utility in assessing exposure to the multitude (tens of thousands) of chemicals representing the reality of exposure. Innovative tools need to be evaluated for their potential contributions to exposure assessment through rapid, cost-efficient methods which allow the simultaneous measurement of multiple chemical agents and gathering of contextual information to inform exposure reduction. These integrated tools and techniques can then be used to refine measurement and predictive modeling methods that support high throughput chemical analysis and exposure assessment.

The proposed research concept represents collaboration between NIEHS (Division of the National Toxicology Program, Division of Intramural Research, and the Clinical Research Unit) and the EPA Office ofResearch and Development (ORD). The partnership includes co- funding with EPA, the sharing of equipment and expertise, and the use of EPA field teams for extensive collection of exposure information.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals born female will be recruited for this study.
* Individuals must be between 35 and 74 years old at the time of enrollment.
* Individuals must be a non-smoker living in a non-smoking home. Individuals who are former smokers or live with a former smoker must be at least one year smoke free at the time of enrollment.
* Individuals must be non-pregnant and non-nursing at the time of enrollment.
* Individuals will not be selected for specific preexisting health conditions but will be excluded if any of the conditions described in Section 5.2 (EXCL 5) are present at the time of enrollment.
* Individuals who spend a majority of their time in the home each day will be recruited for this study. This includes individuals who work from home, are stay-at-home caretakers, retired, unemployed, etc.
* Individuals must use a high number of consumer products. A high consumer product user is someone who uses more than a certain number of products (e.g., 15 or more products a day). This number will be finalized following the completion of a separating screening activity by NIEHS under a separate IRB protocol, and will be defined prior to enrollment of participants in the study.

EXCLUSION CRITERIA:

* Persons born male or female-identifying transgender individuals will be excluded from the study population.
* Individuals younger than 35 years old or older than 74 years old will be excluded from the study population.
* Individuals who smoke, use tobacco products, or any form of electronic cigarettes, personal vaporizers, or electronic nicotine delivery systems will be excluded from the study population. Additionally, based on the pre-screening questionnaire individuals who live in homes with others who use one or more of these products will not be eligible to participate. Prescreening responses will be verified against cotinine test results from Screening Day 1
* Individuals who may be pregnant, are pregnant, or are nursing will be excluded from the study population.
* Individuals with chronic kidney or liver disease or insulin-dependent diabetics based on pre-screening questionnaire will not be eligible to participate in the study.
* Individuals who work outside of the home or spend a majority of their time each day outside of the home for other activities will be excluded from the study population.
* Individuals who use less than a certain number of consumer products (e.g., 15 products per day) will be excluded from the study population.

Ages: 35 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals will be recruited from the RTP area, since they will be required to complete home and clinic visits as part of their study participation.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Primary endpoint will be daily individual exposure estimates for each participant calculated through forward modeling of questionnaire data and environmental measurements and reverse modeling ofbiomarker data. | Ongoing

SECONDARY OUTCOMES:
To evaluate the accuracy of historical consumer product usage questionnaires. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Kyla W Taylor, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-E-0134.html